CLINICAL TRIAL: NCT04662502
Title: Observational, Prospective, Multicentric Study of the Effect of Bifidobacterium Longum 35624 on Quality of Life of Patients With Irritable Bowel Syndrome
Brief Title: Efficacy of Bifidobacterium Longum 35624 on the Quality of Life of IBS Patients With Different Symptom Severity
Status: Completed | Type: Observational
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Other Study IDs: Floravie
Record Dates: First submitted 2020-11-18; First posted 2020-12-10 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Bifidobacterium longum 35624 — Bifidobacterium longum 35624, 1 x 10^9 CFU/capsule, 1 capsule/day over 1 month

SUMMARY:
The main objective of this observatory is to evaluate the effect of Bifidobacterium longum 35624 on the quality of life of IBS patients having different subtypes of transit pattern and different level of symptom severity

DETAILED DESCRIPTION:
This observatory evaluate the effect of Bifidobacterium longum 35624 on the quality of life of IBS patients having different subtypes of transit pattern and different level of symptom severity, after a one-month treatment with Bibidobacterium longum 35624, 1x10^9 CFU/capsule, 1 capsule/day.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age
* Gastroenterology consultation for an Irritable Bowel Syndrome according to Rome IV criteria
* Having received a first prescription of Bifidobacterium longum 35624 during the consultation (independently of participation in the observatory)
* Informed and having declared his/her non-opposition to the study.

Exclusion Criteria:

* Not having a good enough command of reading and comprehension of the French language to correctly complete the questionnaires and the notebook
* Having already taken Bifidobacterium longum 35624
* Having received probiotics or antibiotics within 2 weeks previous
* Having started within the last 7 days a treatment that can interfere with the investigator's evaluation of the investigational product under investigation
* Participant in another trial
* Pregnant or breastfeeding women
* Being under guardianship or curator.
* Not having a good enough command of reading and comprehension of the French language to correctly complete the questionnaires and the notebook

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult outpatients with IBS consulting a gastroenterologist
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Quality of life assessed with the Irritable Bowel Syndrome Quality Of Life questionnaire (IBS-QOL). | Assessed at baseline and after 1 month of treatment
  Change from baseline of quality of life as assessed with the Irritable Bowel Syndrome Quality Of Life questionnaire (IBS-QOL, scoring from 0 to 100, with higher scores indicating better IBS specific quality of life) in IBS patients having different subtypes of transit pattern and different level of symptom severity.

SECONDARY OUTCOMES:
Quality of life subscores assessed with the Irritable Bowel Syndrome Quality Of Life questionnaire (IBS-QOL). | Assessed at baseline and after 1 month of treatment
  Change from baseline of quality of life subscores as assessed with the Irritable Bowel Syndrome Quality Of Life questionnaire (IBS-QOL, scoring from 0 to 100, with higher scores indicating better IBS specific quality of life) in IBS patients having different subtypes of transit pattern and different level of symptom severity.
IBS Symptom Severity | Assessed at baseline and after 1 month of treatment
  Change of IBS Symptom Severity assessed with the IBS Severity Scoring System (IBS-SSS, scoring from 0 to 500, with higher scores indicating worse severity of IBS symptoms)
Change of Stool consistency | Assessed at baseline, day10, day 20 and day 30
  Change of stool consistency assessed with the Bristol stool scale. The Bristol Stool Chart classifies stool according to their shape and consistency and assigns a sample a number from 1-7 depending on its characteristics, corresponding to constipation normal or diarrhea.
Compliance to the treatment | Assessed after 1 month of treatment
  Compliance assessed with patient self-report on a diary
Patient satisfaction | Assessed after 1 month of treatment
  Patient satisfaction with treatment assessed on a 5-point Likert scale, with proposals ranked in ascending order of satisfaction as 1- Not at all satisfied; 2- Unsatisfied; 3- Somewhat satisfied; 4-Satisfied to 5-Very satisfied
Patient's overall impression after treatment | Assessed after 1 month of treatment
  The patient's overall impression of how the product has changed his or her daily activities, symptoms, and quality of life, assessed with the Patients' Global Impression of Change (PGIC) scale. PGIC is a 7-point scale describing patient's rating of overall improvement. Change is rated by patients as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Physician's satisfaction | Assessed after 1 month of treatment
  Physician satisfaction with the treatment for his/her patient assessed on a 5-point Likert scale, with proposals ranked in ascending order of satisfaction as 1- Not at all satisfied; 2- Unsatisfied; 3- Somewhat satisfied; 4-Satisfied to 5-Very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Gyasi K Johnson, PhD, Study Director — Biocodex
Locations (1):
- Hôpital Avicenne, Bobigny, France

IPD SHARING:
Plan to Share IPD: Undecided